CLINICAL TRIAL: NCT01432886
Title: A Phase 1 Study of Eribulin Mesylate With Trastuzumab for Advanced or Recurrent Human Epidermal Growth Factor Receptor 2-Positive (HER2+) Breast Cancer
Brief Title: A Study of Eribulin Mesylate With Trastuzumab for Advanced or Recurrent Human Epidermal Growth Factor Receptor 2-Positive (HER2+) Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-107
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Results first posted 2015-03-30 (Estimated); Last update posted 2016-10-07 (Estimated); Status verified 2016-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — Eribulin mesylate (iv) will be administered on Day 1 and Day 8 of each cycle (3 weeks as 1 cycle). Trastuzumab (iv) will be administered as weekly use or tri-weekly use. Trastuzumab will be administered immediately after eribulin mesylate administration when used concomitantly.

SUMMARY:
The purpose of the study is to evaluate dose limiting toxicity (DLT), investigate the tolerability and safety of eribulin mesylate with trastuzumab combination therapy, and estimate the recommended dose.

ELIGIBILITY:
Inclusion Criteria

* Females aged greater than or equal to 20 years and less than 75 years at the time of informed consent.
* Histologically or cytologically confirmed with breast cancer
* Score 3+ by immunohistochemistry (IHC) or HER2 positive by Fluorescence in Situ Hybridization (FISH) method
* Subjects who meet any of the following criteria:

  * Evidence of recurrence during adjuvant chemotherapy with trastuzumab and taxane
  * Evidence of recurrence within 6 months after adjuvant chemotherapy with trastuzumab and taxane
  * Experienced prior chemotherapy including trastuzumab and taxane for advanced or recurrent breast cancer
* Adequate organ function
* Eastern Cooperative Oncology Group (ECOG)-Performance Status (PS) is 0 or 1
* Subjects who have submitted written informed consent for study entry

Exclusion Criteria

* Subjects with known brain metastasis accompanied by clinical symptoms or requiring active treatment
* Subjects with severe active infection requiring active treatment
* Subjects with large pleural effusions, ascites, or pericardial effusions requiring drainage.
* Hypersensitivity to trastuzumab, halicondrin B or halicondrin B chemical derivatives
* Known positive for human immunodeficiency virus (HIV) test or positive for hepatitis B surface (HBs antigen) or hepatitis C (HCV) by serum test.
* Subjects who are pregnant (positive B-hCG test) or breastfeeding
* Subjects judged to be ineligible for this study by the principal investigator or sub-investigator.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tadashi Nakanishi, Study Director — Eisai Co., Ltd.
Locations (2):
- Japan (2):
  - Kashiwa-shi, Chiba
  - Hidaka-shi, Saitama

REFERENCES:
- [Derived] Mukai H, Saeki T, Shimada K, Naito Y, Matsubara N, Nakanishi T, Obaishi H, Namiki M, Sasaki Y. Phase 1 combination study of eribulin mesylate with trastuzumab for advanced or recurrent human epidermal growth factor receptor 2 positive breast cancer. Invest New Drugs. 2015 Feb;33(1):119-27. doi: 10.1007/s10637-014-0161-y. Epub 2014 Sep 23. PMID 25242374

RESULTS

PARTICIPANT FLOW:
Groups:
- E7389 With Weekly Trastuzumab: Eribulin mesylate (E7389) was administered intravenously on Day 1 and Day 8 of each 3 week cycle. Trastuzumab was administered intravenously weekly, with an initial dose of 4 mg/kg followed by 2 mg/kg for the remaining doses.
- E7389 With Tri-weekly Trastuzumab: Eribulin mesylate (E7389) was administered intravenously on Day 1 and Day 8 of each 3 week cycle. Trastuzumab was administered intravenously tri-weekly, with an initial dose of 8 mg/kg followed by 6 mg/kg for the remaining doses.
Period: Overall Study
Arm/Group | E7389 With Weekly Trastuzumab | E7389 With Tri-weekly Trastuzumab
Started | 6 | 6
Completed | 6 (Discontinuation met per discontinuation criteria) | 6 (Discontinuation met per discontinuation criteria)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E7389 With Weekly Trastuzumab | E7389 With Tri-weekly Trastuzumab | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (5.05) | 49.2 (10.32) | 56.9 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Japanese | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT)
Description: For DLT evaluation, severity (grade) was classified according to common terminology criteria for adverse events version 4.0 (CTCAE v4.0). DLTs were defined as grade 4 neutropenia persisting for more than 7 days; grade 3 or above febrile neutropenia; grade 4 thrombocytopenia or grade 3 thrombocytopenia requiring blood transfusion; non-hematologic toxicity (excluding toxicity related to neutrophils, leukocytes, lymphocytes, platelets, CD4 lymphocytes, anemia, and bone marrow density) greater than or equal to grade 3 (Exceptions: Dose reduction was not required even when the following conditions were met: grade 3 nausea, vomiting, or diarrhea controllable with anti-emetic or anti-diarrheal medication and abnormal laboratory parameter not requiring treatment); and day 8 administration was delayed or skipped as a result of the subject did not meet the dosing riteria within cycle.
Time Frame: Up to 3 weeks
Population: The DLT analysis set included those participants who received at least one dose of study drug and had a DLT assessment in cycle 1 (3 weeks) without deviations from the eribulin mesylate/trastuzumab dosing regimens and other major protocol prescripts. Participants with a DLT, regardless of this criterion, were also included in the DLT analysis set.
Measure: Number; unit: Participants
Arm/Group | E7389 With Weekly Trastuzumab | E7389 With Tri-weekly Trastuzumab
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: The number of subjects who developed 'treatment-emergent adverse events (AEs) and serious adverse events (SAEs) were evaluated.
Time Frame: From signing of informed consent up to 30 days after participant's last treatment dose or up to approximately 2 years
Population: The safety analysis set included all participants who received at least one dose of study drug and had at least one post dose safety evaluation.
Measure: Number; unit: Participants
Groups:
- E7389 With Triweekly Trastuzumab: Eribulin mesylate (E7389) was administered intravenously on Day 1 and Day 8 of each 3 week cycle.
  Trastuzumab was administered intravenously tri-weekly, with an initial dose of 8 mg/kg followed by 6 mg/kg for the remaining doses.
Arm/Group | E7389 With Weekly Trastuzumab | E7389 With Triweekly Trastuzumab
Number analyzed (Participants) | 6 | 6
Participants | 6 | 6

ADVERSE EVENTS:
Time Frame: From signing of informed consent up to 30 days after participant's last treatment dose or up to approximately 2 years
Description: The safety analysis set included all participants who received at least one dose of study drug and had at least one post dose safety evaluation. A subject with two or more treatment emergent adverse events in the same system organ class/preferred term is counted only once for that system organ class/preferred term.
Arm/Group | E7389 With Weekly Trastuzumab | E7389 With Tri-weekly Trastuzumab
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 With Weekly Trastuzumab (N=6) | E7389 With Tri-weekly Trastuzumab (N=6)
Anaemia (Blood and lymphatic system disorders) | 4 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 6 | 6
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 6 | 6
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 2 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Cheilitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Oral dysaesthesia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3
Chest discomfort (General disorders) | 1 | 1
Implant site pain (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 1 | 0
Injection site reaction (General disorders) | 2 | 0
Malaise (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Contrast media reaction (Injury, poisoning and procedural complications) | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 0
Ejection fraction decreased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other